CLINICAL TRIAL: NCT07289438
Title: A Holistic Evaluation of Enneagram Personality Types, Eating Habits, Emotional Eating, Psychological Well-being and Spirituality in Obese Individuals
Brief Title: The Relationship Between Enneagram Personality Types and Eating Behaviors, Emotional Eating, Psychological Well-Being, and Spirituality in Obese Individuals: A Holistic Approach
Acronym: OBEZ-ENNEA
Status: Not yet recruiting | Type: Observational
Sponsor: Diyetisyenin Mutfağı (Other)
Responsible Party: Sponsor
Other Study IDs: OBEZ-ENNEAGRAM-2025
Record Dates: First submitted 2025-06-10; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Obesity; Eating Behavior; Emotional Eating
Keywords: enneagram; personality types; emotional eating; eating habits; psychological well-being; spirituality
MeSH Terms: conditions — Obesity; Feeding Behavior; Emotional Eating; Psychological Well-Being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study explores the relationship between Enneagram personality types and eating behaviors, emotional eating, psychological well-being, and spirituality in obese individuals from a holistic perspective.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 18 and 65 years
* Body Mass Index (BMI) ≥ 30 (classified as obese)
* Literate and able to understand the questionnaire
* Volunteering to participate in the study

Exclusion Criteria:

* Individuals with a current psychiatric diagnosis
* Those who have undergone bariatric surgery in the last year
* Pregnant individuals

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese adult individuals aged 18-65 years, recruited from general population for a study on personality, eating habits, and well-being.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-12-31 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Emotional Eating Score Differences Across Enneagram Personality Types | At baseline (single survey administration)
  To assess whether Emotional Eating Scale scores differ significantly among individuals classified into different Enneagram personality types. Emotional eating will be measured using a validated Emotional Eating Scale, and scores will be compared across personality categories.

SECONDARY OUTCOMES:
Psychological Well-Being Score Differences Across Enneagram Personality Types | At baseline (single survey administration)
  To compare psychological well-being across Enneagram personality types using a validated Psychological Well-Being Scale.
Spirituality Score Differences Across Enneagram Personality Types | At baseline (single survey administration)
  To evaluate differences in spirituality levels across individuals classified into different Enneagram personality types using a validated Spirituality Assessment Instrument.
General Eating Behavior Differences Across Enneagram Personality Types | At baseline (single survey administration)
  To compare general eating behavior patterns across Enneagram personality types using a validated Eating Behavior Questionnaire.
Body Mass Index (BMI) Differences Across Enneagram Personality Types | At baseline (single measurement)
  To determine whether BMI differs across individuals in different Enneagram personality types. BMI will be calculated using measured height and weight.

OTHER OUTCOMES:
Emotional Eating Score Differences Across BMI Categories | At baseline (single survey administration)
  To compare Emotional Eating Scale total scores across BMI categories (normal weight, overweight, obese).
Psychological Well-Being Score Differences Across BMI Categories | At baseline (single survey administration)
  To evaluate whether psychological well-being differs among individuals in different BMI categories.